CLINICAL TRIAL: NCT01559532
Title: Influence of Tourniquet Use and Surgery Duration on the Incidence of Deep Vein Thrombosis in Total Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 222
Record Dates: First submitted 2012-03-13; First posted 2012-03-21 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Deep Vein Thrombosis
Keywords: Deep vein thrombosis; Thromboembolism; Tourniquet; Knee prosthesis.
MeSH Terms: conditions — Venous Thrombosis; Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ATK patients: Patients from our institution that underwent cemented TKA for degenerative knee disorders.

SUMMARY:
This is an observational study to analyze the influence of surgery duration and tourniquet time in the incidence of deep venous thrombosis (DVT) in patients that had undergone total knee arthroplasty (TKA).

DETAILED DESCRIPTION:
Influence of Tourniquet Use and Surgery Duration on the Incidence of Deep Vein Thrombosis in Total Knee Arthroplasty

Tourniquet, Surgery Duration and DVT in TKA.

Abstract:

Objective: The occurrence of deep vein thrombosis (DVT) was evaluated in 78 patients submitted to total knee arthroplasty (TKA), followed by ascending venography (AV), between the seventh and twelfth days postoperative.

Methods: Patients received prophylaxis with oral anticoagulation for 12 days, maintaining INR at around 2.5.

Results: Results showed 45 cases (57.7%) of negative bilateral AV and 33 (42.3%) cases of positivity for DVT. Thirteen cases were of the proximal type DVT, making up 16.7% of the total. We compared the groups with and without DVT, and another which considered only cases with proximal DVT.

Conclusion: The statistical analysis didn't reveal significance in relation to tourniquet time, despite the higher likelihood of proximal DVT after 90 minutes (p=0.08) and surgery duration of more than 120 minutes increases its risk.

Keywords: Deep vein thrombosis. Prophylaxis. Thromboembolism. Tourniquet. Knee prosthesis.

Introduction Total knee arthroplasties (TKAs), together with total hip arthroplasties, are frequently the object of study regarding deep vein thrombosis (DVT) (1); however, DVT also commonly occurs in other knee procedures (2). Despite the importance of this problem and the interest in it, most researchers studying DVT generally focus on prophylaxis for prevention; surprisingly, there have been few studies of the isolated risk factors for DVT associated with TKA. Although there is some controversy about the role of TKA alone as a risk factor for DVT (3-7), some researchers believe that bone manipulation, reaming of the medullary canal, and the duration of the different procedures are relevant risk factors for DVT (8,9). Another important and controversial factor related to TKA is the use of surgical tourniquets. Although all these factors are mentioned in the literature, surgery duration as an isolated risk factor for DVT in TKA has received little attention.

We used ascending venography (AV) to evaluate the association between the use of tourniquets and total procedure duration and the occurrence of DVT during TKA.

Patients and Methods Seventy-eight consecutive patients from our institution underwent cemented TKA for degenerative knee disorders and then underwent AV, for which they gave informed consent, at a point between 7 and 12 days after surgery, after having been discharged from the hospital. Of the 78, 78.2% were women and 21.8% were men, with an average age of 65.1 years (range, 31-88 years; SD, 11.5 years). Osteoarthrosis was the diagnosis in 74.4%, rheumatoid arthritis in 21.8%, and other disorders in 3.8%.

All patients received prophylaxis for DVT with oral anticoagulants for 12 days, with an international normalized ratio being maintained at about 2.5 (range, 2.0-3.0) in all cases. Perioperatively, we recorded total pneumatic tourniquet time and total surgery duration, in minutes. In all cases, the use of a tourniquet was interrupted by hemostasis, after cementation of the implant and before wound closure. Five categories were established for total tourniquet time: <60, 61 to 90, 91 to 120, and >120 minutes. The total procedure duration was defined in the same way; we recorded the times of the initial incision and the last suture stitch made to close the incision. Three categories were defined for procedure duration: <120, 121 to 150, and >150 minutes. Only 2 patients (3.1%) were given a general anesthetic; all the others were given a spinal block.

The study end point was defined as the execution of bilateral AV at a point between 7 and 12 days after surgery, after hospital discharge. The AV was carried out by a specialist in vascular radiology. The technique applied was basically that described by Rabinov and Paulin (10). The presence of clinically manifested DVT and/or pulmonary embolism was also taken in to consideration. The clinical manifestations of DVT were greater edema of the lower limb than would be expected for the procedure, associated with intense pain on palpation of the calf and pain on passive dorsiflexion of the foot.

AV findings were considered positive for DVT in the presence of blood clots in the vein lumens (Figure 1). They were characterized as occurring on the operated side, contralateral or bilateral, and were diagnosed as proximal DVT (more severe) or distal DVT (less severe), depending on the contents of the radiologist's report.

ELIGIBILITY:
Inclusion Criteria:

* patients that underwent cemented total knee arthroplasty

Exclusion Criteria:

* post-operative infection
* inadequate follow-up

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Seventy-eight consecutive patients from our institution underwent cemented TKA for degenerative knee disorders and then underwent AV, for which they gave informed consent, at a point between 7 and 12 days after surgery, after having been discharged from the hospital.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2008-02; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Deep vein thrombosis | 7 days
  Deep vein thrombosis confirmed by ascending venography performed 7 days after total knee arthroplasty.

CONTACTS AND LOCATIONS:
Overall Officials: Arnaldo J Hernandez, Prof. Dr., Study Director — Orthopedics and Traumatology Department - University of Sao Paulo General Hospital
Locations (1):
- Orthopedics Department - University of Sao Paulo General Hospital, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Bergqvist D, Bergentz SE, Fredin H. Thromboembolism in orthopaedic surgery. Acta Orthop Scand. 1984 Jun;55(3):247-50. doi: 10.3109/17453678408992348. No abstract available. PMID 6204500
- [Background] Stringer MD, Steadman CA, Hedges AR, Thomas EM, Morley TR, Kakkar VV. Deep vein thrombosis after elective knee surgery. An incidence study in 312 patients. J Bone Joint Surg Br. 1989 May;71(3):492-7. doi: 10.1302/0301-620X.71B3.2785998.
- [Background] Caprini JA, Arcelus JI, Reyna JJ. Effective risk stratification of surgical and nonsurgical patients for venous thromboembolic disease. Semin Hematol. 2001 Apr;38(2 Suppl 5):12-9. doi: 10.1016/s0037-1963(01)90094-0. PMID 11449339
- [Background] Geerts WH, Heit JA, Clagett GP, Pineo GF, Colwell CW, Anderson FA Jr, Wheeler HB. Prevention of venous thromboembolism. Chest. 2001 Jan;119(1 Suppl):132S-175S. doi: 10.1378/chest.119.1_suppl.132s. No abstract available. PMID 11157647
- [Background] Haas S. Prevention of venous thromboembolism: recommendations based on the International Consensus and the American College of Chest Physicians Sixth Consensus Conference on Antithrombotic Therapy. Clin Appl Thromb Hemost. 2001 Jul;7(3):171-7. doi: 10.1177/107602960100700301. PMID 11441977
- [Background] Stulberg BN, Insall JN, Williams GW, Ghelman B. Deep-vein thrombosis following total knee replacement. An analysis of six hundred and thirty-eight arthroplasties. J Bone Joint Surg Am. 1984 Feb;66(2):194-201. PMID 6693445
- [Background] Kim YH, Kim VE. Factors leading to low incidence of deep vein thrombosis after cementless and cemented total knee arthroplasty. Clin Orthop Relat Res. 1991 Dec;(273):119-24. PMID 1959258
- [Background] Haas S. Managing the risk of venous thromboembolism in orthopedics: concluding remarks. Orthopedics. 1997 Feb;20 Suppl:26-7. No abstract available. PMID 9048405
- [Background] Zaw HM, Osborne IC, Pettit PN, Cohen AT. Risk factors for venous thromboembolism in orthopedic surgery. Isr Med Assoc J. 2002 Nov;4(11):1040-2. No abstract available. PMID 12489502
- [Background] Rabinov K, Paulin S. Roentgen diagnosis of venous thrombosis in the leg. Arch Surg. 1972 Feb;104(2):134-44. doi: 10.1001/archsurg.1972.04180020014004. No abstract available. PMID 5008903
- [Background] Brookenthal KR, Freedman KB, Lotke PA, Fitzgerald RH, Lonner JH. A meta-analysis of thromboembolic prophylaxis in total knee arthroplasty. J Arthroplasty. 2001 Apr;16(3):293-300. doi: 10.1054/arth.2001.21499. PMID 11307125
- [Background] Freedman KB, Brookenthal KR, Fitzgerald RH Jr, Williams S, Lonner JH. A meta-analysis of thromboembolic prophylaxis following elective total hip arthroplasty. J Bone Joint Surg Am. 2000 Jul;82-A(7):929-38. doi: 10.2106/00004623-200007000-00004. PMID 10901307
- [Background] Lotke PA, Ecker ML, Alavi A, Berkowitz H. Indications for the treatment of deep venous thrombosis following total knee replacement. J Bone Joint Surg Am. 1984 Feb;66(2):202-8. PMID 6693446
- [Background] Wauke K, Nagashima M, Kato N, Ogawa R, Yoshino S. Comparative study between thromboembolism and total knee arthroplasty with or without tourniquet in rheumatoid arthritis patients. Arch Orthop Trauma Surg. 2002 Nov;122(8):442-6. doi: 10.1007/s00402-002-0404-9. Epub 2002 Apr 18. PMID 12442180
- [Background] Wakankar HM, Nicholl JE, Koka R, D'Arcy JC. The tourniquet in total knee arthroplasty. A prospective, randomised study. J Bone Joint Surg Br. 1999 Jan;81(1):30-3. doi: 10.1302/0301-620x.81b1.8971. PMID 10067997